CLINICAL TRIAL: NCT03626506
Title: Evaluation of spironolactoNe Versus Indapamide on Target Organ Damage in Patients With Obesity and hYpertension(ENVOY)
Brief Title: Spironolactone Versus Indapamide in Obese and Hypertensive Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: University of Michigan (Other); Peking University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMUJI007
Record Dates: First submitted 2018-08-03; First posted 2018-08-13 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-04

CONDITIONS: Hypertension
Keywords: spironolactone; Indapamide; Obesity; Hypertension; Target organ damage
MeSH Terms: conditions — Hypertension; Obesity | interventions — Spironolactone; Indapamide; Amlodipine

STUDY DESIGN:
Intervention Model Description: randomized, controlled, open-label trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- spironolactone (Experimental): Subjects will take spironolactone 20~40mg once daily on top of amlodipine 5~10mg once daily.
  Interventions: Drug: Spironolactone; Drug: Amlodipine
- indapamide (Active Comparator): Subjects will take indapamide 1.5~3.0mg once daily on top of amlodipine 5~10mg once daily.
  Interventions: Drug: Indapamide; Drug: Amlodipine

INTERVENTIONS:
Drug: Spironolactone — After a 2-week run-in period on amlodipine, patients who still have SBP ≥ 140mmHg will take spironolactone 20mg once daily on top of amlodipine for 12 months. During the first two months after randomization, spironolactone can be titrated to 40mg if office SBP remains ≥ 140mmHg.
  Arms: spironolactone
Drug: Indapamide — After a 2-week run-in period on amlodipine, patients who still have SBP ≥ 140mmHg will take extended-release indapamide 1.5mg once daily on top of amlodipine for 12 months. During the first two months after randomization, indapamide can be titrated to 3mg if office SBP remains ≥ 140mmHg.
  Arms: indapamide
Drug: Amlodipine — After a 2-week run-in period on amlodipine 5mg once daily, patients who still have SBP ≥ 140mmHg will be randomized to add spironolactone 20mg once daily or extended-release indapamide 1.5mg once daily to amlodipine for 12 months. During the first two months after randomization, amlodipine can be titrated to 10mg if office SBP remains ≥ 140mmHg.

SUMMARY:
Most recent guidelines continue to recommend thiazide diuretics as first-line agents for patients with hypertension in spite of the potential metabolic side effects, while mineralocorticoid receptor antagonists (MRAs), such as spironolactone or eplerenone, are mainly recommended to be used in patients with resistant hypertension or heart failure.However,animal studies demonstrated that MRAs induce beneficial changes in left ventricular remodeling and prevent or partially reverse cardiac fibrosis and pathological hypertrophy that contribute to the development of diastolic heart failure. MRAs have also been shown to decrease inflammation and myocardial fibrosis in patients with obesity and the metabolic syndrome. In the proposed study, the investigators planned to randomize 400 patients with essential hypertension and increased waist circumference to receive spironolactone or indapamide in combination with amlodipine for 12 months. The effects of the two diuretics on target organ damage detected by changes in left atrial volume index(LAVI) by echocardiography reflecting left ventricular diastolic dysfunction or changes in carotid-femoral pulse wave velocity(PWV) reflecting arterial stiffness will be compared. The potential role of MRAs as initial therapy for patients with essential hypertension and visceral obesity will be evaluated.

DETAILED DESCRIPTION:
Thiazide diuretics have been widely used for the management of essential hypertension, especially in patients with salt-sensitive hypertension. Most recent guidelines continue to recommend thiazide diuretics as first-line agents for all patients with hypertension in spite of the potential metabolic side effects such as hypokalemia, hypertriglyceridemia, impaired glucose tolerance and increases in serum cholesterol and uric acid. However, mineralocorticoid receptor antagonists (MRAs), such as spironolactone or eplerenone, are mainly recommended to be used in patients with resistant hypertension or heart failure because they have never been evaluated for efficacy in reducing cardiovascular events in uncomplicated patients with hypertension. Indeed, it has been demonstrated that MRAs reduced total mortality or cardiovascular death in patients with systolic heart failure with severe or mild symptoms and in patients undergoing hemodialysis for chronic renal dysfunction. Animal studies demonstrated that MRAs induce beneficial changes in left ventricular remodeling and prevent or partially reverse cardiac fibrosis and pathological hypertrophy that contribute to the development of diastolic heart failure. MRAs have also been shown to decrease inflammation and myocardial fibrosis in patients with obesity and the metabolic syndrome. Of interest is the recent finding in EMPHASIS-HF study in which almost all of the benefit of eplerenone was found in those patients with an increased waist circumference. Therefore, the investigators have reason to believe that MRAs will be more effective than thiazide diuretics in preventing target organ damage and can be used initially in patients with essential hypertension and visceral obesity. In the proposed study, the investigators planned to randomize 400 patients with essential hypertension and increased waist circumference to receive spironolactone or indapamide in combination with amlodipine for 12 months. The effects of the two diuretics on target organ damage detected by changes in left atrial volume index(LAVI) by echocardiography reflecting left ventricular diastolic dysfunction or changes in carotid-femoral pulse wave velocity(PWV) reflecting arterial stiffness will be compared. If it proves that spironolactone as first-line antihypertensive medication is more effective than indapamide in target organ protection, the investigators would propose a large scale cardiovascular outcome trial to evaluate cardiovascular events in patients with essential hypertension and visceral obesity.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with essential hypertension aged between 18-80years
2. Office systolic blood pressure (SBP)≥140mmHg and <180mmHg without treatment or on one antihypertensive drug or SBP<140mmHg on two antihypertensive drugs
3. Waist circumference ≥90cm for males, ≥ 80cm for females

Exclusion Criteria:

1. Secondary hypertension.
2. Symptomatic congestive heart failure or history of heart failure.
3. History of ischemic stroke, unstable angina or myocardial infarction;
4. Atrial fibrillation
5. Serum creatinine ≥ 2.0mg/dl or eGFR≤ 30 ml/min/1.73 m2
6. Serum K+ ≥ 5.0 mmol/L or ≤3.5 mmol/L

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2019-02-13 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
left atrial volume index (LAVI) | 12 months
  change in left atrial volume index (LAVI) from baseline to the end of study period of 12 months

SECONDARY OUTCOMES:
carotid-femoral pulse wave velocity (PWV) | 12 months
  change in carotid-femoral pulse wave velocity (PWV) from baseline to the end of study period of 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Wang Guisong, MD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China